CLINICAL TRIAL: NCT00217243
Title: Evoked (Magnetic) Cortical Fields for the Comparative Study of Mechanisms Underlying Chronic Non-malignant Pain in Peripheral Nerve Injury (CRPS II) and CRPS I (Chronic Regional Pain Syndrome I)
Brief Title: Evoked Fields After Median and Ulnar Stimulation
Status: Completed | Type: Observational
Sponsor: Medical Center Alkmaar (Other)
Collaborators: Rudolf Magnus Institute - University of Utrecht (Other); Technical University of Twente (Other); VU University of Amsterdam (Other); Dept. of Clinical Neurophysiology - VU University Hospital Amsterdam (Other); Human Brain Mapping and Cortical Imaging Laboratory, Centre for Sensory - Motor Interaction, (Unknown); Aalborg University (Other)
Responsible Party: P.J. Theuvenet, anesthesiologist, Medical Center Alkmaar, The Netherlands
Other Study IDs: NH04-196
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Complex Regional Pain Syndromes
Keywords: Pain; Magnetoencephalography; Median; Ulnar; Causalgia; Complex regional pain syndrome; Evoked fields; Nerve injury; Neuropathic pain
MeSH Terms: conditions — Complex Regional Pain Syndromes; Pain; Causalgia; Neuralgia | interventions — Lidocaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pain study Netherlands: 20 healthy subjects 20 patients with a traumatic unilateral peripheral nerve injury 20 patients with CRPS I
  Interventions: Other: Evoked fields before and after a local block (Xylocaine)

INTERVENTIONS:
Other: Evoked fields before and after a local block (Xylocaine) — MEG registration after electrical median and ulnar nerve stimulation in subjects and patients. In the patient group another MEG was performed after an anaesthetic block (1-2 ml Lidocaine 1%) at the site of the nerve injury producing a painfree state
  Other Names: All subjects were rated with the HC code, 1 to 20; All patients with nerve injury were rated with the A - code, 1 to 20; All patients with CRPS I were rated with the C - code, 1 to 20

SUMMARY:
In order to be able to study the effects of evoked fields with magnetoencephalography (MEG) in two groups of patients, comparison is made with a group of healthy volunteers.

DETAILED DESCRIPTION:
This study is directed at the (central and / or peripheral) mechanisms of pain and the cortical changes (plasticity) due to chronic non-malignant pain in two groups of patients and one healthy volunteer group.

The aim of the study is further to evaluate cortical processes by MEG (and fMRI, if feasible) to quantify and qualify the responses, localise the generators and study the effects of a pain therapy.

To search for patterns that may result in diagnostic criteria and have an indicative value for the treatment and the monitoring of the effects.

Finally the study not only intends to support clinical diagnosis but also to provide tools to monitor treatment and support the choice (algorithm) between SCS and SAN. An algorithm, facilitating decision making between these two treatments, will be promoted. It should also provide a clinical decision tool for the use of SAN

ELIGIBILITY:
Inclusion Criteria:

CRPS I:

* (Absolute) functio laesa, secondary pain and cold sensations
* (Relative) abnormal skin colour, allodynia, hyperalgesia, hyperpathia, hyperhydrosis,oedema, increased nail growth, increased hair growth. (At least 4 need to be present).

CRPS II:

* All the previous but evidence of traumatic peripheral nerve injury.

Exclusion Criteria:

* General condition
* Pregnancy
* Technical implants (pacemaker, SCS: disturbs MEG)

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: subjetcs were sampled from the hospital staff of two hospitals all patients were recruited from one hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-06; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Theuvenet, MD, Principal Investigator — Medical Center Alkmaar
Locations (1):
- Medical Center of Alkmaar, Alkmaar, North Holland, Netherlands

REFERENCES:
- [Background] Theuvenet PJ, Dunajski Z, Peters MJ, van Ree JM. Responses to median and tibial nerve stimulation in patients with chronic neuropathic pain. Brain Topogr. 1999 Summer;11(4):305-13. doi: 10.1023/a:1022210704505. PMID 10449261
- [Result] Theuvenet PJ, van Dijk BW, Peters MJ, van Ree JM, Lopes da Silva FL, Chen AC. Whole-head MEG analysis of cortical spatial organization from unilateral stimulation of median nerve in both hands: no complete hemispheric homology. Neuroimage. 2005 Nov 1;28(2):314-25. doi: 10.1016/j.neuroimage.2005.06.010. Epub 2005 Jul 22. PMID 16040256
- [Result] Theuvenet PJ, van Dijk BW, Peters MJ, van Ree JM, Lopes da Silva FL, Chen AC. Cortical characterization and inter-dipole distance between unilateral median versus ulnar nerve stimulation of both hands in MEG. Brain Topogr. 2006 Winter;19(1-2):29-42. doi: 10.1007/s10548-006-0010-1. PMID 16977490